CLINICAL TRIAL: NCT03796533
Title: Pharmacokinetics Variability of Posaconazole (PCZ) and Its Glucuronide Metabolite During Induction and Consolidation Treatments in Patients With Acute Myeloid Leukemia (AML): a Covariate Analysis With the Tablets Formulation and Evaluation of the Potential Risk of Hepatotoxicity
Acronym: Posa-Pk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL18_0429; 2018-003488-67 (Other: ID-RCB)
Record Dates: First submitted 2018-11-16; First posted 2019-01-08 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML-PCZ-UGT1A4 gene
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Posaconazole pharmacokinetics (Other): Patients with AML over the age of 18 years treated with intensive chemotherapy in induction and consolidation whose was under antifungal prophylaxis by PCZ formulation tablets.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — * PCZ will be used as recommended in tablet formulation at an initial dosage of 300 mg twice a day on the first day and then once a day at a dose of 300 mg the following days.
  * PCZ prophylaxis will be started on the same day as the start of chemotherapy and will be continued until the end of aplasia.
  * The dosage of the PCZ can be adjusted according to the results of the PCZ assay. It may be interrupted if the transaminase level is greater than 3 times higher than normal (3N) or on medical decision.
  Other Names: PCZ

SUMMARY:
Among its authorized indications, posaconazole (PCZ) is prescribed for prophylaxis in onco-hematology patients at high risk of invasive fungal infections. This azole antifungal has a low bioavailability. The enteric-coated tablets form available since mid-2015 has significantly improved its pharmacokinetic profile compared to the oral suspension form initially used. According to the recommendations of The European Conference on Infections in Leukemia (ECIL-6), the minimum serum concentration desirable for prophylaxis is 0.7 mg/L. This concentration threshold was difficult to achieve in onco-hematology patients treated with oral suspension.

The investigators retrospectively collected and analyzed 201 results of residual PCZ serum concentrations from 91 onco-hematology patients on Noxafil® tablets prophylaxis. The median concentration of PCZ was 1.08 mg/L. In this study, the pharmacokinetics of tablet-PCZ showed significant inter-individual variability. Thus, while 25% of the concentrations remained below the recommended threshold of 0.7 mg/L (25% percentile = 0.69 mg/L), exposure to PCZ was greater than 2.63 mg/L in 10% of cases. This level of exposure, however, did not have obvious hepatic repercussions. Nevertheless, further studies involving larger cohorts are needed to clarify a hypothetical relationship between serum PCZ concentration and the occurrence of hepatic toxicity.

In addition, the investigators found significant intra-individual variability in PCZ exposure (CV = 48.8%), especially in leukemic patients. This variability is probably related to a modification during the treatment of the physio-pathological conditions of the patient likely to impact the pharmacokinetics of PCZ (absorption, distribution, metabolism, etc.) as well as the effect of possible pharmacokinetic drug interactions.

The metabolism of PCZ is mediated primarily by the uridine diphosphate (UDP)-glucuronosyltransferase 1A4 (UGT1A4) pathway. Although hepatic metabolism of PCZ is low compared with other azoles (such as itraconazole or voriconazole), differences in the metabolic capacity of UGT1A4 may alter PCZ exposure. A previous study of the oral suspension form had shown that low concentrations of PCZ were associated with a high ratio of PCZ-glucuronide / PCZ concentrations. Two genetic variants of the gene encoding UGT1A4 are associated with a decrease in the metabolic clearance of glucuronide drugs via UGT1A4. A recent study suggests less exposure to PCZ in the presence of UGT1A4 polymorphism.

The main objective of the investigator's project is to study prospectively in a homogeneous population of patients treated by intensive chemotherapy for acute myeloid leukemia (induction and consolidation) the pharmacokinetics of PCZ administered in its tablet formulation, and in particular:

* Clinical and biological tolerance of high concentrations of PCZ
* The influence of clinical and demographic covariates on PCZ and PCZ-glucuronide ratio
* The influence of genetic variants of UGT1A4 on PCZ metabolism (PCZ-glucuronide / PCZ ratio).

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 or over
2. Patients with AML de novo or secondary to myelodysplastic syndrome or therapy-related AML except acute myeloid leukemia (AML3)
3. Patient hospitalized for the treatment of leukemia (induction chemotherapy or consolidation)
4. General state retained (ECOG performance scale ≤ 3)
5. alanine aminotransferase aspartate transaminase (ASAT) and alanine aminotransferase (ALAT) ≤ 2.5 times the upper limit of normal (ULN), total bilirubin ≤ 2 times the ULN, creatinine <150 μmol / L unless these biological abnormalities are related to leukemia
6. Patients affiliated or beneficiaries of a social security scheme (Social Security or Universal Medical Coverage)
7. Having read and understood the information sheet and signed the informed consent

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia (AML3)
2. History of uncontrolled cancer for at least two years
3. Patient included in another clinical study that may interfere with the objectives of this study
4. Treatment with antifungal other than posaconazole
5. Severe uncontrolled infection at the time of inclusion
6. Positive serology for HIV 1 or 2 or human T-cell lymphoma virus (HTLV 1) or 2, or active viral infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
7. Pregnant woman (beta positive HCG) or breastfeeding
8. A woman of childbearing potential who can not justify the use of effective contraception during treatment with Noxafil®
9. Patient incapacitated, under guardianship, curators or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Evolution of the blood concentration of posaconazole and its metabolite from the beginning of treatment to the end of the induction phase (pharmacokinetic). | Day 21
  Posaconazole (PCZ) treatment will start at Day 1 at the beginning of induction/ consolidation therapy.
  * For the pharmacokinetics study of PCZ during induction, blood samples (5 mL) will be taken on days 3, 7, 14 and 21. Predoses (just prior to a daily dose) or trough concentrations (C0) will be collected on days 3, 7, 14 and 21. A peak concentration (at 3 hours post dose) will also be collected on day 14.
  * After achieving complete remission, patients receive a consolidation cure. During the consolidation cures, trough concentrations will be collected on days 3, 7, 14 and 21. A peak concentration (at 3 hours post dose) will also be collected on day 14.

SECONDARY OUTCOMES:
Search and identification by sequencing gene variants of UGT1A4 | At diagnosis
  The blood sample (5 mL) for the study of polymorphisms of the UGT1A4 gene will be performed before the initiation of induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Hematology department, Pierre-Bénite, France

REFERENCES:
- [Derived] Parant F, Gagnieu MC, Di-Pilla L, Deloire A, Joassard A, Millet A, Barthelemy D, Payen L, Ducastelle-Lepretre S. Impact of UGT1A4 Polymorphisms on the Posaconazole Serum Trough Concentrations in Patients With Acute Myeloid Leukemia Receiving Delayed-Release Tablets. Ther Drug Monit. 2025 Oct 1;47(5):609-618. doi: 10.1097/FTD.0000000000001319. Epub 2025 Mar 4. PMID 40044655